CLINICAL TRIAL: NCT04390594
Title: Multicentre, Open Label, Randomised, Adaptative Clinical Trial of Efficacy and Safety of Treatment Regimens in Adult COVID-19 Patients in Senegal
Brief Title: Efficacy and Safety Evaluation of Treatment Regimens in Adult COVID-19 Patients in Senegal
Acronym: SEN-CoV-Fadj
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: In conclusion, the results of the SEN-CoV Fadj trial to date do not meet the objectives of the clinical trial and the sample size required to meet them is clearly too large to be achieved within a reasonable time.
Sponsor: Institut Pasteur de Dakar (Other)
Collaborators: Fann Hospital, Senegal (Unknown); Ministry of Health, Senegal (Other Government); Diamniadio Children Hospital, Senegal (Unknown); Dalal Jamm Hospital, Senegal (Other); Institut Pasteur Korea (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2020-002
Record Dates: First submitted 2020-05-14; First posted 2020-05-15 (Actual); Last update posted 2024-06-21 (Actual); Status verified 2020-09

CONDITIONS: COVID-19
Keywords: COVID-19; SARS-CoV-2; Efficacy; Safety; Senegal; Nafamostat mesilate
MeSH Terms: conditions — COVID-19 | interventions — nafamostat

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of Care (No Intervention): The Standard of Care is the treatment which is the most adapted to the patient in the clinician's opinion. It could include the combination of Hydroxychloroquine and Azithromycin in the absence of contraindication.
- Standard of Care + Nafamostat mesilate (Experimental): * The Standard of Care is the treatment which is the most adapted to the patient in the clinician's opinion. It could include the combination of Hydroxychloroquine and Azithromycin in the absence of contraindication.
  * Nafamostat mesilate
  Interventions: Drug: Nafamostat Mesilate

INTERVENTIONS:
Drug: Nafamostat Mesilate — Nafamostat mesilate continuous intravenous injection. Daily dose ranging between 0.1 mg/kg/h and 0.2 mg/kg/h, based on the severity and underlying disease of the clinical trial participant.
  Administration for 10-14 days based on the severity and underlying disease of the clinical trial participant
  Arms: Standard of Care + Nafamostat mesilate

SUMMARY:
COVID-19 is an emerging pandemic disease affecting most countries including Senegal, caused by the new coronavirus (SARS-CoV-2) which was first detected in the city of Wuhan in China in December 2019. A rapid spread of the disease has occurred at a global scale, associated with a mortality rate of 3.4%. The first case in Africa was declared on February 15, 2020 in Egypt and the first case in Senegal was declared on March 2nd, 2020.

In this context, the SEN-CoV-Fadj clinical trial aims to evaluate efficacy and safety, among adults, of different therapeutic regimens considered optimal according to current knowledge, as well as available and adapted to Sub-Saharan Africa. This trial is nested into a cohort of confirmed cases of COVID-19 in Senegal aiming to understand the main clinical, biological, virologic and immunological characteristics of the infection. The protocol of the cohort is based and adapted from the International Severe Acute Respiratory and Emerging Infection Consortium (ISARIC) / World Health Organization (WHO) Clinical Characterisation Protocol (CCP).

The Nafamostat mesilate, whose antiviral, anticoagulant an anti-inflammatory activities have been shown, has been eligible for SEN-CoV-Fadj for the treatment of moderate to severe COVID-19 cases.

DETAILED DESCRIPTION:
COVID-19 is an emerging pandemic disease affecting most countries including Senegal, caused by the new coronavirus (SARS-CoV-2) which was first detected in the city of Wuhan in China in December 2019. A rapid spread of the disease has occurred at a global scale, associated with a mortality rate of 3.4%. The first case in Africa was declared on February 15, 2020 in Egypt and the first case in Senegal was declared on March 2nd, 2020.

In this context, the SEN-CoV-Fadj clinical trial aims to evaluate efficacy and tolerance, among adults, of different therapeutic options considered optimal according to current knowledge, as well as available and adapted to Sub-Saharan Africa. This trial is nested into a cohort of confirmed cases of COVID-19 in Senegal aiming to understand the main clinical, biological, virologic and immunological characteristics of the infection. The protocol of the cohort is based and adapted from the International Severe Acute Respiratory and Emerging Infection Consortium (ISARIC) / World Health Organization (WHO) Clinical Characterisation Protocol (CCP).

The Nafamostat mesilate, whose antiviral, anticoagulant an anti-inflammatory activities have been shown, has been eligible for SEN-CoV-Fadj for the treatment of moderate to severe COVID-19 cases. Its efficacy and safety will be evaluated against the standard of care used in Senegal.

The primary objective is to :

Evaluate and compare viral clearance between the different therapeutic interventions.

The secondary objectives are to:

* Evaluate and compare efficacy of the different therapeutic regimens
* Evaluate and compare the tolerance of the different therapeutic regimens
* Evaluate and compare the impact of the different therapeutic interventions on the length of hospitalization and other clinical measurements

ELIGIBILITY:
Inclusion Criteria:

* Confirmed cases of SARS-CoV-2 infection hospitalized in reference services identified by the Ministry of Health and Social Action of Senegal
* Adults (≥18 years)
* Full understanding and consent to participate to the trial
* No contraindications to taking the tested treatments
* Clinical status from 3 to 5 on the seven-category ordinal scale
* Pneumonia highlighted by infiltration of the lungs by chest CT scan or chest radiography
* Absence of contraindications to radiographic examinations (X-ray and/or CT scan) for diagnosis and/or follow-up
* Inclusion in the 72 hours following the radiological pneumonia confirmation

Non-inclusion Criteria:

* Pregnant or breastfeeding woman
* Patient at high risk of death within 3 days of inclusion, in the clinician's opinion
* Corrected QT interval (QTc) >500ms
* Heart electrical dysfunction: atrioventricular block Mobitz type II second-degree, high-grade or complete without a functioning pacemaker
* Uncontrolled and clinically significant heart diseases, such as arrhythmia, angina or decompensated congestive heart failure
* Kidney failure (Cl < 30 mL/min)
* Patients with liver cirrhosis whose Child-Puch score is B or C
* Patients who have liver disease abnormalities with ALT or AST > 5 times ULN
* Patients who have a known HIV status
* Patients who have other clinically-important diseases in decompensation which may interfere with the evaluation or completion of the tested treatment's procedure, in the clinician's opinion
* Patients with a clinical or psychological condition which, in the clinician's opinion, does not allow adequate evaluation of the tested treatment
* Known allergy to the studied treatment regimen
* Other contraindications with the studied treatment regimen
* Known drug-drug interaction with a treatment usually taken by the participant contraindicating one of the studied treatment regimen

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2020-08-13 (Actual); Primary Completion 2023-02-08 (Actual); Study Completion 2023-02-08 (Actual)

PRIMARY OUTCOMES:
SARS-CoV-2 viral load level | Day 7
  Real time-PCR (RT-PCR) result of the naso- and oro-pharyngeal sample

SECONDARY OUTCOMES:
Vital status | Day 15
Proportion of patients with serious adverse events reported during the clinical trial. | through study completion, an average of 7 months
Length of hospitalization | through hospitalization, an average of 2 weeks
Length of hospitalization in a resuscitation unit | through hospitalization, an average of 2 weeks
Duration of oxygen therapy | through hospitalization, an average of 2 weeks
Maximum quick SOFA (qSOFA) score during hospitalisation | through hospitalization, an average of 2 weeks
Clinical status on the seven-category ordinal scale | through hospitalization, an average of 2 weeks
  1. not hospitalized with resumption of normal activities;
  2. not hospitalized, but unable to resume normal activities;
  3. hospitalization, not requiring supplemental oxygen;
  4. hospitalization, requiring supplemental oxygen;
  5. hospitalization, requiring nasal high-flow oxygen therapy and/or noninvasive mechanical ventilation;
  6. hospitalization, requiring extracorporeal membrane oxygenation and/or invasive mechanical ventilation;
  7. death.

CONTACTS AND LOCATIONS:
Overall Officials: Moussa Seydi, MD, Principal Investigator — Fann Hospital, Senegal; Amadou A. Sall, PhD, Study Director — Institut Pasteur de Dakar, Senegal; Fabien Taieb, MD, PhD, Principal Investigator — Institut Pasteur de Dakar, Senegal
Locations (3):
- Senegal (3):
  - Infectious and Tropical Diseases Department, Fann Hospital, Dakar
  - Diamniadio Children Hospital, Diamniadio
  - Dalal Jamm Hospital, Guédiawaye

IPD SHARING:
Plan to Share IPD: Undecided